CLINICAL TRIAL: NCT03294642
Title: Ingestion of Potatoes as a Nutritional Strategy to Improve Cycling Time-trial Performance in Endurance Trained Cyclists
Brief Title: Potato Ingestion and Time-trial Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Alliance for Potato Research and Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 18104
Record Dates: First submitted 2017-09-19; First posted 2017-09-27 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2017-09

CONDITIONS: Exercise Performance
Keywords: exercise; FODMAP; gastrointestinal; endurance; cycling
MeSH Terms: conditions — Motor Activity | interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Trial 1 (Experimental): Water Intervention: In one of the 3 cycling trials, participants will receive only water and no carbohydrate supplementation during the 2 hour cycling challenge.
  Interventions: Dietary Supplement: Water
- Trial 2 (Experimental): Carbohydrate Gel Intervention: In one of the 3 cycling trials, participants will receive carbohydrate supplementation in the form of commercially available gels (15g every 15 minutes) during the 2 hour cycling challenge.
  Interventions: Dietary Supplement: Carbohydrate Gel
- Trial 3 (Experimental): Potatoes Intervention: In one of the 3 cycling trials, participants will receive carbohydrate supplementation in the form of pureed russet potato (15g every 15 minutes) during the 2 hour cycling challenge.
  Interventions: Dietary Supplement: Potatoes

INTERVENTIONS:
Dietary Supplement: Potatoes — Pureed russet potatoes will be used as a carbohydrate supplement for participants during one of the three cycling challenges.
  Arms: Trial 3
Dietary Supplement: Carbohydrate Gel — Commercially available PowerBar PowerGel will be used for the carbohydrate gel condition during one of the three cycling challenges.
  Arms: Trial 2
Dietary Supplement: Water — Water will be used as a control during one of the three cycling challenges (participants will not receive any carbohydrate supplementation).
  Other Names: Control
  Arms: Trial 1

SUMMARY:
This research study evaluates the feasibility and appropriateness of potatoes as an ergogenic aid in comparison to the currently promoted sports gels during a cycling challenge and time trial. Using a crossover design, trained cyclists will complete three separate cycling challenges and subsequent time trials in which they will consume either potatoes, commercially available sports gels, or water only.

DETAILED DESCRIPTION:
The metabolic demands created by endurance activities, which include muscle and liver glycogen depletion as well as losses in body fluids and electrolytes, are significant limitations to the performance potential of the athlete. For this reason, a well-supported recommendation exists for such athletes to consume a carbohydrate formula, in particular, one containing electrolytes during their activity.

Currently, most commercially available exercise-nutrition products for use in endurance activities come at relatively high costs to the athlete. Moreover, the ingredients used within this market vary and could therefore hinder their effectiveness. For example, Fermentable Oligosaccharides Disaccharides Monosaccharides and Polyols (FODMAPs) potentially present in common sports foods (i.e. excess fructose) are known to alter gastrointestinal (GI) function in some individuals. Indeed, 25-70% of endurance athletes experience GI symptoms during exercise. Given the prevalence of exercise induced GI discomfort in this population, it is possible that GI symptoms limit the adherence to nutritional recommendations during exercise. Therefore identification of a targeted nutrition strategy that maximizes GI effectiveness and dietary adherence is warranted.

An alternative to the commercially available sports foods are whole foods. Specifically, white potatoes, which have a high GI index, indicates that their carbohydrate content is readily available. Additionally, potatoes naturally contain potassium, an important electrolyte. Because of these characteristics, potatoes provide the potential to be a low-cost alternative, and merit investigation. To this point, we know of no studies that have explored the effectiveness of white potatoes as an ergogenic aid. Therefore, the purpose of this study is to examine how capable potatoes are at off-setting the losses in muscle and liver glycogen and electrolytes compared to the current products available on the market, i.e. "sports gels."

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* ≥150 km/wk of cycling mileage
* ≥6 months of prior training history
* VO2peak values ≥45 ml/kg/min for females and ≥50 ml/kg/min for males
* Aged between 20-40 years

Exclusion Criteria:

* Chronic Smoking or tobacco use
* Active cardiovascular disease
* Diabetes Mellitus or other metabolic disorders
* Liver kidney, or urinary disease
* Musculoskeletal/Orthopedic disorders (e.g., osteoarthritis, rheumatoid arthritis, tendinitis, gout, fibromyalgia, patellar tendinopathy, or chronic low back pain)
* Neuromuscular disorders
* hypertension
* Diagnosed GI tract diseases
* Heart Disease
* Bleeding or clotting disorders
* Neurological disease
* Epilepsy
* Respiratory disease
* Pregnancy
* Contraindications for exercise
* <150 km/wk of cycling mileage
* <6 months of prior training history
* VO2peak values <45 ml/kg/min for females and <50 ml/kg/min for males

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2019-09-29 (Actual); Study Completion 2019-09-29 (Actual)

PRIMARY OUTCOMES:
Time trial performance measured in minutes | 1 year
  Comparison of time trial performance times between potatoes and sports gel conditions to determine effectiveness of potatoes as an ergogenic aid.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas A Burd, Ph.D, Principal Investigator — University of Illinois at Urbana-Champaign, Department of Kinesiology
Locations (1):
- Freer Hall, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No